CLINICAL TRIAL: NCT07349641
Title: Tirzepatide With Progestin Intrauterine Device to Treat Endometrial Hyperplasia and Grade 1 Endometrial Cancer in Overweight and Obese Women
Brief Title: A Study of Weight Loss Intervention With Tirzepatide and Progestin Intrauterine Device to Treat Endometrial Hyperplasia and Grade 1 Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2026-00081; NCI-2026-00081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MDA24-19-01 (Other: M D Anderson Cancer Center); MDA24-19-01 (Other: DCP); P30CA016672 (NIH); UG1CA242609 (NIH)
Record Dates: First submitted 2026-01-16; First posted 2026-01-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Atypical Hyperplasia/Endometrioid Intraepithelial Neoplasia; FIGO Grade 1 Endometrial Endometrioid Adenocarcinoma
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Specimen Handling; X-Rays; Dilatation and Curettage; Magnetic Resonance Spectroscopy; Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (LNG-IUD, tirzepatide) (Experimental): Patients undergo LNG-IUD placement at baseline or on day 0 and then receive tirzepatide SC QW for 26 weeks in the absence of disease progression or unacceptable toxicity. Patients who qualify for tirzepatide or another weight loss medication as determined by primary provider may continue to receive treatment beyond 26 weeks as per standard of care. Additionally, patients undergo cervical culture sample collection, chest x-ray, and MRI or CT with transvaginal ultrasound during screening and blood sample collection and EMB throughout the study. Patients may also undergo D&C during screening.
  Interventions: Procedure: Biospecimen Collection; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Dilation and Curettage; Procedure: Endometrial Biopsy; Procedure: Magnetic Resonance Imaging; Other: Medical Device Usage and Evaluation; Drug: Tirzepatide; Procedure: Transvaginal Ultrasound

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo cervical culture and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Dilation and Curettage — Undergo D&C
  Other Names: D and C; D&C; dilatation and curettage; Dilation and Curettage of the Uterus; Dilation and Curettage Procedure
Procedure: Endometrial Biopsy — Undergo EMB
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Medical Device Usage and Evaluation — Undergo LNG-IUD placement
Drug: Tirzepatide — Given SC
Procedure: Transvaginal Ultrasound — Undergo transvaginal ultrasound
  Other Names: transvaginal sonography; TVS; TVU

SUMMARY:
This phase II trial studies whether adding tirzepatide injections to a levonorgestrel intrauterine device (LNG-IUD) improves pathologic response (absence of cancer cells in tissue samples after treatment) in women with endometrial atypical hyperplasia/endometrial intraepithelial neoplasia (AH/EIN) or grade 1 endometrial cancer who are overweight or obese. Endometrial cancer occurrence has continued to rise in the United States. Over half of endometrial cancer cases are thought to be attributable to being overweight and obese, and the risk relationship appears to be weight dependent. AH/EIN is a precancerous condition of the endometrium (the uterus or womb) where the lining of the uterus grows abnormally thick, and the cells become abnormal. Women with this thickening have a higher-than-average risk of developing endometrial cancer if left untreated. The usual approach for patients who have AH/EIN and grade 1 endometrial cancer is the removal of the uterus. While surgical treatment is generally safe and effective, it may not be the best approach for some patients. Tirzepatide injections are a type of glucagon-like peptide 1 (GLP-1) agonist which have been shown to drive weight loss. The LNG-IUD is a small, T-shaped device inserted into the uterus that releases the hormone levonorgestrel. Levonorgestrel is being studied in the prevention of endometrial cancer. Adding tirzepatide injections to LNG-IUD may help overweight or obese women with AH-EIN or grade 1 endometrial cancer lose weight, which may improve pathologic response.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the proportion of pathological complete response (pCR) on endometrial biopsy (EMB) at 26 weeks among patients receiving combined treatment with tirzepatide (dosed weekly) and levonorgestrel intrauterine device (LNG-IUD) for management of endometrial atypical hyperplasia/endometrial intraepithelial neoplasia (AH/EIN) and grade 1 endometrioid endometrial cancer in overweight or obese women compared to historical controls who received LNG-IUD alone.

SECONDARY OBJECTIVES:

I. To determine the proportion of participants who achieve sustained pathologic complete response on EMB at 52 weeks (12 months) compared to historical controls.

II. To estimate the time to complete response and duration of response, up to 52 weeks (12 months) compared to historical controls.

III. To determine the rate of hyperplasia persistence and progression to endometrial cancer at 26 and 52 weeks (6 and 12 months) compared to historical controls.

IV. To estimate percent change in cell proliferation (Ki-67+) at 12, 26, 39 and 52 weeks compared to historical controls and baseline.

V. To estimate percent change in hemoglobin A1C (HbA1C) at 12, 26, 39 and 52 weeks compared to baseline.

VI. To estimate percent weight change every 4 weeks up to week 20 and then at weeks 26, 39 and 52 compared to baseline.

VII. To estimate percent change in fasting blood glucose every 4 weeks up to week 20 and then at weeks 26, 39, and 52 compared to baseline.

EXPLORATORY OBJECTIVES:

I. To investigate the effect of GLP-1 agonism on the endometrial immune microenvironment at 12, 26, 39 and 52 weeks compared to baseline.

II. To investigate the effect of GLP-1 agonism on systemic inflammation and metabolic markers at 12 26, 39 and 52 weeks compared to baseline.

III. To investigate weight independent effects of GLP-1 agonism on cell proliferation (Ki-67+) at 12, 26, 39 and 52 weeks compared to baseline.

IV. To investigate the effect of tirzepatide and LNG-IUD on treatment response based on molecular ProMisE (Proactive Molecular Risk Classifier for Endometrial Cancer) classification at 26 and 52 weeks.

OUTLINE:

Patients undergo LNG-IUD placement at baseline or on day 0 and then receive tirzepatide subcutaneously (SC) once a week (QW) for 26 weeks in the absence of disease progression or unacceptable toxicity. Patients who qualify for tirzepatide or another weight loss medication as determined by primary provider may continue to receive treatment beyond 26 weeks as per standard of care. Additionally, patients undergo cervical culture sample collection, chest x-ray, and magnetic resonance imaging (MRI) or computed tomography (CT) with transvaginal ultrasound during screening and blood sample collection and EMB throughout the study. Patients may also undergo dilation and curettage (D&C) during screening.

After completion of study treatment, patients are followed up at weeks 30, 39, and 52.

ELIGIBILITY:
Inclusion Criteria:

* Women who have a pathologic diagnosis of AH/EIN or grade 1 endometrioid endometrial cancer confirmed on dilation and curettage (D&C) and desire non-surgical management, who are overweight (body mass index [BMI] ≥ 27 kg/m^2) with a weight-related comorbidity (hypertension, type 2 diabetes, or high cholesterol) or obese (BMI ≥ 30 kg/m^2) with or without weight-related comorbidities
* Prior progesterone treatment for conditions other than AH/EIN or endometrial cancer is allowed, but a 28-day washout period is required before levonorgestrel IUD placement. If archival tissue is available from prior to any progesterone treatment but after the diagnosis of AH/EIN/EC, the washout period is not needed
* Age ≥ 18 years. Because no dosing or adverse event (AE) data are currently available on the use of tirzepatide in participants < 18 years of age, children and adolescents < 18 years of age are excluded from this study but will be eligible for future pediatric trials, if applicable
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For participants with a history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load
* Participants on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible
* Ability to comply with EMB every 3 months
* Women currently using oral hypoglycemic agents (e.g., metformin) are eligible for the study
* Ability to understand and the willingness to sign a written informed consent document in English or Spanish

Exclusion Criteria:

* Women with grade 2-3 endometrioid, or women with serous, clear cell, mucinous, squamous, transitional cell, sarcomas, or carcinosarcoma histology
* Evidence of extrauterine spread of disease on imaging or during surgical evaluation
* Participants may not be receiving any other investigational agents or anticancer therapies (including chemotherapy, radiation therapy, hormonal, or antibody-based therapy). Prior treatment should have a minimum washout period of 14 days
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the levonorgestrel IUD or any GLP-1 agonist
* Uncontrolled intercurrent illness, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study. Because of this, a pregnancy test is part of the screening for the study and women who are pregnant or planning pregnancy within 6 months after the end of the study will be excluded. The LNG-IUD is an Food and Drug Administration (FDA)-approved contraceptive agent. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.

Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with tirzepatide, breastfeeding should be discontinued if the mother is treated with tirzepatide

* Women who have any severe and/or uncontrolled medical conditions such as:

  * Unstable angina pectoris, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease,
  * Symptomatic congestive heart failure of New York Heart Association class III or IV,
  * Active (acute or chronic) or uncontrolled severe infection (not responding to antibiotics), liver diseases such as cirrhosis and decompensated liver disease,
  * Known severely impaired lung function (spirometry and diffusion capacity of the lung for carbon monoxide [DLCO] 50% or less of normal and oxygen [O2] saturation 88% or less at rest on room air), or
  * Active, bleeding diathesis
* Other malignancies within the past 3 years except for basal or squamous cell carcinoma of the skin
* Active (acute or chronic) or uncontrolled severe infections (not responding to antibiotics), including acute pelvic inflammatory disease
* Congenital or acquired uterine anomaly which distorts the uterine cavity
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use one additional highly effective method of contraception in addition to the LNG-IUD during the study and 8 weeks after. Acceptable highly effective contraception methods include a combination of any of the following:

  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
  * Total abstinence or;
  * Male sterilization;
  * Female bilateral tubal ligation or bilateral salpingectomy Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy or tubal ligation at least six weeks prior to study initiation. When the diagnosis of menopause is unclear based on patient history, we will assess follicle-stimulating hormone \ (FSH) levels for confirmation. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential
* Tirzepatide is contraindicated in patients with a personal or family history of medullary thyroid carcinoma (MTC) or in patients with multiple endocrine neoplasia (MEN) 2A or 2B. Such women will be excluded
* Participants taking any other prescription medication intended to induce weight loss (i.e., orlistat, phentermine-topiramate, naltrexone-bupropion). A 28-day washout period is required if such women want to enter the study
* Participants on active intermittent fasting
* Participants currently using insulin for glucose control
* Participants who have previously used any glucagon-like peptide (GLP) medications (liraglutide, semaglutide, dulaglutide, exenatide), whether oral or injectable
* Participants diagnosed with Lynch Syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-07-06 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Weighted pathological complete response (pCR) | At 26 weeks
  The weighted pCR is weighted by the prevalence of endometrial atypical hyperplasia (AH) and endometrioid endometrial cancer (EC) in the reference group. The reference group is the historical control reported by Westin et al. The prevalence of the AH group was 63% and was 37% for the EC group in the study. Will be calculated with its 95% confidence interval. The stratified pCR rates for AH and EC will also be reported separately, along with their 95% confidence intervals.

SECONDARY OUTCOMES:
Proportion of participants who achieve pCR on endometrial biopsy | At 52 weeks
  Will be compared to historical controls. Will be calculated with 95% confidence intervals.
Time to complete response and duration of response | Up to 52 weeks
  The time will be measured in months and estimated using the Kaplan-Meier method. Will be compared to historical controls. The log-rank test may be applied to evaluate differences in time-to-event outcomes between different prognostic groups. Cox proportional hazards regression will be employed, when possible, to further evaluate the effects of important covariates on time-to-event outcomes, adjusting for clinical and demographic characteristics of interest (e.g., age, race, tobacco use).
Rate of hyperplasia persistence and progression to EC | At 26 and 52 weeks
  Will be compared to historical controls as assessed by standard pathologic criteria. Will be calculated with 95% confidence intervals.
Percent change in cell proliferation | At baseline and 12, 26, 39, and 52 weeks
  Will assess anti-Ki67 primary antibody (Dakopatts) within pre-treatment biopsy and post-treatment biopsies. Will also compare with historical controls. Will summarize percent changes from baseline using mean, standard deviation, median and range. Graphical tools may be used to visualize changes in continuous variables over time.
Percent change in hemoglobin A1C | At baseline and weeks 12, 26, 39, and 52
  Will be measured by means of commercially available assays. Will summarize percent changes from baseline using mean, standard deviation, median and range. Graphical tools may be used to visualize changes in continuous variables over time.
Percent weight change | Every 4 weeks up to week 20 and at weeks 26, 39, and 52
  Will summarize percent changes from baseline using mean, standard deviation, median and range. Graphical tools may be used to visualize changes in continuous variables over time. Paired t-tests or Wilcoxon signed-rank tests will be used to compare weight changes at different time points and to assess weight independent effects.
Percent change in fasting blood glucose | Every 4 weeks up to week 20 and at weeks 26, 39, and 52
  Will summarize percent changes from baseline using mean, standard deviation, median and range. Graphical tools may be used to visualize changes in continuous variables over time.

OTHER OUTCOMES:
Change in the endometrial immune microenvironment | At baseline and 12, 26, 39, and 52 weeks
  Changes pre- and post-treatment will be assessed using paired t-tests or Wilcoxon signed-rank tests. Analyses will be stratified by diabetes status (different inflammatory profile than nondiabetics) and by weight loss (to assess weight loss-independent effects), and if necessary, reasons for non-surgery (those who wish to avoid surgery to preserve fertility versus [vs.] those who are not candidates for surgery).
Change in systemic inflammation and metabolic markers | At baseline and 12, 26, 39 and 52 weeks
  Will summarize percent changes from baseline using mean, standard deviation, median and range. Graphical tools may be used to visualize changes in continuous variables over time. Changes pre- and post-treatment will be assessed using paired t-tests or Wilcoxon signed-rank tests. Analyses will be stratified by diabetes status (different inflammatory profile than nondiabetics) and by weight loss (to assess weight loss-independent effects), and if necessary, reasons for non-surgery (those who wish to avoid surgery to preserve fertility vs. those who are not candidates for surgery).
Weight-independent effects of glucagon-like peptide 1 on cell proliferation (Ki-67+) | At baseline and 12, 26, 39 and 52 weeks
Effect of intervention on treatment response | At 26 and 52 weeks
  Will evaluate the effect of the intervention (combined treatment of tirzepatide and levonorgestrel intrauterine device) on treatment response stratified by Proactive Molecular Risk Classifier for Endometrial Cancer classification.

CONTACTS AND LOCATIONS:
Overall Officials: Roni N Wilke, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm